CLINICAL TRIAL: NCT04136392
Title: The Global cVAD Study
Acronym: cVAD
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Abiomed Inc. (Industry)
Collaborators: Beth Israel Deaconess Medical Center (Other); Yale University (Other)
Responsible Party: Sponsor
Other Study IDs: cVAD; USPella (Other: Abiomed, Inc.); The Global cVAD Registry (Other: Abiomed, Inc.)
Record Dates: First submitted 2019-10-09; First posted 2019-10-23 (Actual); Last update posted 2021-05-10 (Actual); Status verified 2021-05

CONDITIONS: Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Eligible Patients: The population to be enrolled in this study includes patients whose intended treatment is to receive mechanical circulatory support with the ABIOMED, Inc. hemodynamic support devices per the treating physician's discretion and best practices.
  Interventions: Device: ABIOMED, Inc. hemodynamic support devices

INTERVENTIONS:
Device: ABIOMED, Inc. hemodynamic support devices — ABIOMED, Inc. hemodynamic support technology are the smallest and least invasive percutaneous ventricular support blood pumps available on the market. They are routinely used in clinical practice in a variety of clinical scenarios to support patients in prophylactic or emergent settings.

SUMMARY:
The intent of the Global cVAD Study is to utilize observational data of the ABIOMED, Inc. hemodynamic support devices in real-world settings to drive best practice usage patterns identified through study analysis, to serve as a tool to measure and improve the quality of patient care and to serve as a resource for future research and regulatory filings.

DETAILED DESCRIPTION:
Ongoing, observational, multicenter, records review of patients receiving the ABIOMED, Inc. hemodynamic support device(s). To collect in-hospital data, a waiver of consent and authorization will be requested to avoid significant biases in data reporting due to the extremely high mortality. To collect the post-discharge data on subjects who survive the index hospitalization, an informed consent will be obtained from those subjects or a waiver of informed consent will be used to collect data if the subject was implanted greater than a year from enrollment. Data will be collected through the review of existing medical records and subject telephone interview. Clinical follow-up as an office visit is not required for this study protocol. However, clinical follow-up and event-driven visits (e.g. re-hospitalizations) may occur as clinically warranted. At each follow-up time point, a telephone call to the subject will be attempted to obtain updated medical history and self-assessed cardiac function. In addition to the telephone call, the subject's medical records at the study site will be reviewed for cardiac-related clinic visits and/or cardiac-related re-hospitalization, including echocardiographic imaging. All data collected for this study will be reported on study specific electronic Case Report Forms (eCRFs) and entered into a controlled 21CFRPart11 compliant Electronic Data Capture (EDC) System by the designee at the participating site. Monitoring of the study data will be performed according to the study monitoring plan. Monitoring may be performed on-site or remotely and will not be conducted by anyone involved in data collection. A Clinical Events Committee (CEC) may be formed by the Sponsor. If convened, the CEC, an independent adjudication body composed of cardiologists and cardiac surgeons will adjudicate whether the site-reported adverse events and/or MACCE meet the study definitions for these events, and the relatedness of the events to the procedure and the device. A Steering Committee composed of internationally recognized investigators and experts in the field of interventional cardiology, cardiovascular surgery, cardiac electrophysiology, heart failure and mechanical circulatory support was established to provide technical and scientific oversight of the study.

ELIGIBILITY:
Inclusion Criteria:

1. All subjects in the study population are eligible for enrollment at the time of receiving support from an ABIOMED, Inc. hemodynamic support device, or at the time of attempt to implant an ABIOMED, Inc. hemodynamic support device.

Exclusion Criteria:

1. Patients in whom an attempt to implant an ABIOMED, Inc. hemodynamic support device did not occur.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects who received mechanical circulatory support with an ABIOMED, Inc. hemodynamic support device per treating physician's discretion and best practices will be considered eligible for enrollment. Subjects in whom an attempt was made to implant an ABIOMED, Inc. hemodynamic support device will also be included, even though the attempt was unsuccessful. An attempt is defined as the ABIOMED, Inc. hemodynamic support catheter came in contact with the subject's skin but was not successfully placed.
Sampling Method: Non-Probability Sample
Enrollment: 20000 (Estimated)
Dates: Start 2017-07-14 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events including Major Adverse Cardiac and Cerebrovascular Events | January 2025
  Incidence of Adverse Events including Major Adverse Cardiac and Cerebrovascular Events measured through site-reported events in study EDC through anticipatory primary completion date of January 2025.

CONTACTS AND LOCATIONS:
Overall Officials: Ali Almedhychy, MD, Study Director — Abiomed Inc.
Locations (51):
- United States (51):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Banner Health Research Institute, Banner Good Samaritan Hospital, Phoenix, Arizona
  - Banner University Medical Center, Tucson, Arizona
  - University of Southern California Keck Hospital, Los Angeles, California
  - Cedars Sinai, Los Angeles, California
  - Hoag Memorial Hospital Presbyterian, Newport Beach, California
  - The Center for Advanced Research Excellence - Delray Medical Center, Delray Beach, Florida
  - St. Vincent's Medical Center, Jacksonville, Florida
  - Mercy Hospital Research Institute, Miami, Florida
  - University of Miami, Miami, Florida
  - Orlando Health, Orlando, Florida
  - University Cardiology Associates, Augusta, Georgia
  - WellStar Research Institute, Marietta, Georgia
  - University of Kansas Hospital, Kansas City, Kansas
  - University of Louisville School of Medicine, Louisville, Kentucky
  - Tulane University Medical Center, New Orleans, Louisiana
  - Ochsner Clinic Health Services Corporation, New Orleans, Louisiana
  - Tufts Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital - Corrigan Minehan Heart Center, Boston, Massachusetts
  - St. Vincent Hospital, Worcester, Massachusetts
  - University of Michigan Cardiovascular Center, Ann Arbor, Michigan
  - Detroit Medical Center, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Ascension St. John Hospital, Detroit, Michigan
  - Spectrum Health, Grand Rapids, Michigan
  - Beaumont Health Center, Royal Oak, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - St. Luke's Hospital, Kansas City, Missouri
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Northwell Health, Manhasset, New York
  - Winthrop University Hospital, Mineola, New York
  - Icahn School of Medicine at Mt. Sinai, New York, New York
  - Columbia University Medical Center, New York, New York
  - Mercy Health Anderson, Cincinnati, Ohio
  - University Hospital Cleveland Medical Center, Cleveland, Ohio
  - Good Samaritan Hospital, Dayton, Ohio
  - Mercy Health - Fairfield Hospital Research Center, Fairfield, Ohio
  - Integris Cardiovascular Physicians, Oklahoma City, Oklahoma
  - Albert Einstein Medical Center, Philadelphia, Pennsylvania
  - Pinnacle Health Cardiovascular Institute Inc., Wormleysburg, Pennsylvania
  - Jackson General Hospital, Jackson, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Baylor Heart and Vascular Institute, Dallas, Texas
  - Plaza Medical Center of Fort Worth, Fort Worth, Texas
  - Baylor College of Medicine - TX Heart Institute, Houston, Texas
  - The University of Texas - Health Science Center & Medical School at Houston, Houston, Texas
  - Virginia Commonwealth University Health System, Richmond, Virginia
  - Carilion Medical Center, Roanoke, Virginia
  - University of Washington, Seattle, Washington
  - Charleston Area Medical Center, Charleston, West Virginia
  - West Virginia University Hospital, Morgantown, West Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Seyfarth M, Sibbing D, Bauer I, Frohlich G, Bott-Flugel L, Byrne R, Dirschinger J, Kastrati A, Schomig A. A randomized clinical trial to evaluate the safety and efficacy of a percutaneous left ventricular assist device versus intra-aortic balloon pumping for treatment of cardiogenic shock caused by myocardial infarction. J Am Coll Cardiol. 2008 Nov 4;52(19):1584-8. doi: 10.1016/j.jacc.2008.05.065. PMID 19007597
- [Background] Dixon SR, Henriques JP, Mauri L, Sjauw K, Civitello A, Kar B, Loyalka P, Resnic FS, Teirstein P, Makkar R, Palacios IF, Collins M, Moses J, Benali K, O'Neill WW. A prospective feasibility trial investigating the use of the Impella 2.5 system in patients undergoing high-risk percutaneous coronary intervention (The PROTECT I Trial): initial U.S. experience. JACC Cardiovasc Interv. 2009 Feb;2(2):91-6. doi: 10.1016/j.jcin.2008.11.005. PMID 19463408
- [Background] O'Neill WW, Kleiman NS, Moses J, Henriques JP, Dixon S, Massaro J, Palacios I, Maini B, Mulukutla S, Dzavik V, Popma J, Douglas PS, Ohman M. A prospective, randomized clinical trial of hemodynamic support with Impella 2.5 versus intra-aortic balloon pump in patients undergoing high-risk percutaneous coronary intervention: the PROTECT II study. Circulation. 2012 Oct 2;126(14):1717-27. doi: 10.1161/CIRCULATIONAHA.112.098194. Epub 2012 Aug 30. PMID 22935569
- [Background] Griffith BP, Anderson MB, Samuels LE, Pae WE Jr, Naka Y, Frazier OH. The RECOVER I: a multicenter prospective study of Impella 5.0/LD for postcardiotomy circulatory support. J Thorac Cardiovasc Surg. 2013 Feb;145(2):548-54. doi: 10.1016/j.jtcvs.2012.01.067. Epub 2012 Mar 9. PMID 22405676
- [Background] Anderson MB, Goldstein J, Milano C, Morris LD, Kormos RL, Bhama J, Kapur NK, Bansal A, Garcia J, Baker JN, Silvestry S, Holman WL, Douglas PS, O'Neill W. Benefits of a novel percutaneous ventricular assist device for right heart failure: The prospective RECOVER RIGHT study of the Impella RP device. J Heart Lung Transplant. 2015 Dec;34(12):1549-60. doi: 10.1016/j.healun.2015.08.018. Epub 2015 Sep 8. PMID 26681124
- [Background] Dangas GD, Kini AS, Sharma SK, Henriques JP, Claessen BE, Dixon SR, Massaro JM, Palacios I, Popma JJ, Ohman M, Stone GW, O'Neill WW. Impact of hemodynamic support with Impella 2.5 versus intra-aortic balloon pump on prognostically important clinical outcomes in patients undergoing high-risk percutaneous coronary intervention (from the PROTECT II randomized trial). Am J Cardiol. 2014 Jan 15;113(2):222-8. doi: 10.1016/j.amjcard.2013.09.008. PMID 24527505
- [Background] Kovacic JC, Kini A, Banerjee S, Dangas G, Massaro J, Mehran R, Popma J, O'Neill WW, Sharma SK. Patients with 3-vessel coronary artery disease and impaired ventricular function undergoing PCI with Impella 2.5 hemodynamic support have improved 90-day outcomes compared to intra-aortic balloon pump: a sub-study of the PROTECT II trial. J Interv Cardiol. 2015 Feb;28(1):32-40. doi: 10.1111/joic.12166. PMID 25689546
- [Background] Cohen MG, Ghatak A, Kleiman NS, Naidu SS, Massaro JM, Kirtane AJ, Moses J, Magnus Ohman E, Dzavik V, Palacios IF, Heldman AW, Popma JJ, O'Neill WW. Optimizing rotational atherectomy in high-risk percutaneous coronary interventions: insights from the PROTECT IotaIota study. Catheter Cardiovasc Interv. 2014 Jun 1;83(7):1057-64. doi: 10.1002/ccd.25277. Epub 2013 Nov 18. PMID 24174321
- [Background] Sjauw KD, Konorza T, Erbel R, Danna PL, Viecca M, Minden HH, Butter C, Engstrom T, Hassager C, Machado FP, Pedrazzini G, Wagner DR, Schamberger R, Kerber S, Mathey DG, Schofer J, Engstrom AE, Henriques JP. Supported high-risk percutaneous coronary intervention with the Impella 2.5 device the Europella registry. J Am Coll Cardiol. 2009 Dec 15;54(25):2430-4. doi: 10.1016/j.jacc.2009.09.018. PMID 20082934
- [Background] O'Neill WW, Schreiber T, Wohns DH, Rihal C, Naidu SS, Civitello AB, Dixon SR, Massaro JM, Maini B, Ohman EM. The current use of Impella 2.5 in acute myocardial infarction complicated by cardiogenic shock: results from the USpella Registry. J Interv Cardiol. 2014 Feb;27(1):1-11. doi: 10.1111/joic.12080. Epub 2013 Dec 13. PMID 24329756
- [Background] Cohen MG, Matthews R, Maini B, Dixon S, Vetrovec G, Wohns D, Palacios I, Popma J, Ohman EM, Schreiber T, O'Neill WW. Percutaneous left ventricular assist device for high-risk percutaneous coronary interventions: Real-world versus clinical trial experience. Am Heart J. 2015 Nov;170(5):872-9. doi: 10.1016/j.ahj.2015.08.009. Epub 2015 Aug 15. PMID 26542494
- [Background] Lemaire A, Anderson MB, Lee LY, Scholz P, Prendergast T, Goodman A, Lozano AM, Spotnitz A, Batsides G. The Impella device for acute mechanical circulatory support in patients in cardiogenic shock. Ann Thorac Surg. 2014 Jan;97(1):133-8. doi: 10.1016/j.athoracsur.2013.07.053. Epub 2013 Oct 1. PMID 24090575
- [Background] Valgimigli M, Steendijk P, Sianos G, Onderwater E, Serruys PW. Left ventricular unloading and concomitant total cardiac output increase by the use of percutaneous Impella Recover LP 2.5 assist device during high-risk coronary intervention. Catheter Cardiovasc Interv. 2005 Jun;65(2):263-7. doi: 10.1002/ccd.20380. PMID 15895406
- [Background] Remmelink M, Sjauw KD, Henriques JP, de Winter RJ, Vis MM, Koch KT, Paulus WJ, de Mol BA, Tijssen JG, Piek JJ, Baan J Jr. Effects of mechanical left ventricular unloading by Impella on left ventricular dynamics in high-risk and primary percutaneous coronary intervention patients. Catheter Cardiovasc Interv. 2010 Feb 1;75(2):187-94. doi: 10.1002/ccd.22263. PMID 19941329
- [Background] Kawashima D, Gojo S, Nishimura T, Itoda Y, Kitahori K, Motomura N, Morota T, Murakami A, Takamoto S, Kyo S, Ono M. Left ventricular mechanical support with Impella provides more ventricular unloading in heart failure than extracorporeal membrane oxygenation. ASAIO J. 2011 May-Jun;57(3):169-76. doi: 10.1097/MAT.0b013e31820e121c. PMID 21317769
- [Background] Meyns B, Stolinski J, Leunens V, Verbeken E, Flameng W. Left ventricular support by catheter-mounted axial flow pump reduces infarct size. J Am Coll Cardiol. 2003 Apr 2;41(7):1087-95. doi: 10.1016/s0735-1097(03)00084-6. PMID 12679206
- [Background] Naidu SS. Novel percutaneous cardiac assist devices: the science of and indications for hemodynamic support. Circulation. 2011 Feb 8;123(5):533-43. doi: 10.1161/CIRCULATIONAHA.110.945055. No abstract available. PMID 21300961
- [Background] Burkhoff D, Naidu SS. The science behind percutaneous hemodynamic support: a review and comparison of support strategies. Catheter Cardiovasc Interv. 2012 Nov 1;80(5):816-29. doi: 10.1002/ccd.24421. Epub 2012 Apr 18. PMID 22431494
- [Background] Remmelink M, Sjauw KD, Henriques JP, de Winter RJ, Koch KT, van der Schaaf RJ, Vis MM, Tijssen JG, Piek JJ, Baan J Jr. Effects of left ventricular unloading by Impella recover LP2.5 on coronary hemodynamics. Catheter Cardiovasc Interv. 2007 Oct 1;70(4):532-7. doi: 10.1002/ccd.21160. PMID 17896398
- [Background] Cotter G, Williams SG, Vered Z, Tan LB. Role of cardiac power in heart failure. Curr Opin Cardiol. 2003 May;18(3):215-22. doi: 10.1097/00001573-200305000-00007. PMID 12826823
- [Background] Fincke R, Hochman JS, Lowe AM, Menon V, Slater JN, Webb JG, LeJemtel TH, Cotter G; SHOCK Investigators. Cardiac power is the strongest hemodynamic correlate of mortality in cardiogenic shock: a report from the SHOCK trial registry. J Am Coll Cardiol. 2004 Jul 21;44(2):340-8. doi: 10.1016/j.jacc.2004.03.060. PMID 15261929
- [Background] Torgersen C, Schmittinger CA, Wagner S, Ulmer H, Takala J, Jakob SM, Dunser MW. Hemodynamic variables and mortality in cardiogenic shock: a retrospective cohort study. Crit Care. 2009;13(5):R157. doi: 10.1186/cc8114. Epub 2009 Oct 2. PMID 19799772
- [Background] Mendoza DD, Cooper HA, Panza JA. Cardiac power output predicts mortality across a broad spectrum of patients with acute cardiac disease. Am Heart J. 2007 Mar;153(3):366-70. doi: 10.1016/j.ahj.2006.11.014. PMID 17307413
- [Background] Sauren LD, Accord RE, Hamzeh K, de Jong M, van der Nagel T, van der Veen FH, Maessen JG. Combined Impella and intra-aortic balloon pump support to improve both ventricular unloading and coronary blood flow for myocardial recovery: an experimental study. Artif Organs. 2007 Nov;31(11):839-42. doi: 10.1111/j.1525-1594.2007.00477.x. PMID 18001394
- [Background] Reesink KD, Dekker AL, Van Ommen V, Soemers C, Geskes GG, van der Veen FH, Maessen JG. Miniature intracardiac assist device provides more effective cardiac unloading and circulatory support during severe left heart failure than intraaortic balloon pumping. Chest. 2004 Sep;126(3):896-902. doi: 10.1378/chest.126.3.896. PMID 15364772
- [Background] Henriques JP, Ouweneel DM, Naidu SS, Palacios IF, Popma J, Ohman EM, O'Neill WW. Evaluating the learning curve in the prospective Randomized Clinical Trial of hemodynamic support with Impella 2.5 versus Intra-Aortic Balloon Pump in patients undergoing high-risk percutaneous coronary intervention: a prespecified subanalysis of the PROTECT II study. Am Heart J. 2014 Apr;167(4):472-479.e5. doi: 10.1016/j.ahj.2013.12.018. Epub 2014 Jan 3. PMID 24655695
- [Derived] Velagapudi P, Bellumkonda L, Cohen DJ, Lansky AJ, Abu-Much A, Thompson JB, Schonning MJ, Redfors B, Zhou Z, Grines CL, Maini AS, Li Y, Batchelor WB, O'Neill WW. Clinical outcomes of aortic stenosis patients undergoing Impella-supported high-risk percutaneous coronary intervention. Front Cardiovasc Med. 2026 Jan 7;12:1638259. doi: 10.3389/fcvm.2025.1638259. eCollection 2025. PMID 41573507
- [Derived] Lemor A, Shah T, Thompson JB, Protty MB, Mamas MA, Kinnaird T, Bharadwaj AS, Truesdell AG, Schonning MJ, Zhang Y, Hussain Y, Falah B, Cohen DJ, Redfors B, Baron SJ, Witzke CF, Dixon SR, Basir MB, Lansky AJ, O'Neill WW. Novel risk score for patients undergoing Impella-assisted high-risk percutaneous coronary intervention. Cardiovasc Revasc Med. 2025 Dec;81:86-94. doi: 10.1016/j.carrev.2025.05.031. Epub 2025 May 30. PMID 40541479
- [Derived] Maini AS, Abu-Much A, Redfors B, Wollmuth JR, Basir MB, Faraz HA, Thompson JB, Schonning MJ, Falah B, Moses JW, O'Neill WW. Outcomes among patients with coronary bifurcation lesions undergoing Impella-supported high-risk percutaneous coronary intervention. Am Heart J. 2025 Dec;290:6-16. doi: 10.1016/j.ahj.2025.05.013. Epub 2025 May 22. PMID 40412495
- [Derived] Bonnet G, Rommel KP, Falah B, Lansky AJ, Zhang Y, Schonning MJ, Redfors B, Burkhoff D, Cohen DJ, Basir MB, O'Neill WW, Granada JF. Impact of Mean Blood Pressure Profiles in Percutaneous Left Ventricular Assist Device-Supported High-Risk Percutaneous Coronary Intervention: The PROTECT III Study. J Am Heart Assoc. 2025 May 20;14(10):e036367. doi: 10.1161/JAHA.124.036367. Epub 2025 May 15. PMID 40371603
- [Derived] Jakob P, Lansky AJ, Basir MB, Schonning MJ, Falah B, Zhou Z, Batchelor WB, Abu-Much A, Grines CL, O'Neill WW, Stahli BE. Characteristics and Outcomes of Older Patients Undergoing Protected Percutaneous Coronary Intervention With Impella. J Am Heart Assoc. 2025 May 6;14(9):e038509. doi: 10.1161/JAHA.124.038509. Epub 2025 Apr 16. PMID 40240978
- [Derived] Abu-Much A, Grines CL, Chen S, Batchelor WB, Zhao D, Falah B, Maini AS, Redfors B, Bellumkonda L, Bharadwaj AS, Moses JW, Truesdell AG, Zhang Y, Zhou Z, Baron SJ, Lansky AJ, Basir MB, O'Neill WW, Cohen DJ. Clinical outcomes among patients with mitral valve regurgitation undergoing Impella-supported high-risk PCI. Int J Cardiol. 2024 Dec 15;417:132555. doi: 10.1016/j.ijcard.2024.132555. Epub 2024 Sep 11. PMID 39270940
- [Derived] Falah B, Redfors B, Zhao D, Bharadwaj AS, Basir MB, Thompson JB, Patel RAG, Schonning MJ, Abu-Much A, Zhang Y, Batchelor WB, Grines CL, O'Neill WW. Implications of anemia in patients undergoing PCI with Impella-support: insights from the PROTECT III study. Front Cardiovasc Med. 2024 Jul 18;11:1429900. doi: 10.3389/fcvm.2024.1429900. eCollection 2024. PMID 39091353
- [Derived] Bharadwaj AS, Abu-Much A, Maini AS, Zhou Z, Li Y, Batchelor WB, Grines CL, Baron SJ, Redfors B, Lansky AJ, Basir MB, O'Neill WW. Angiographic Characteristics and Clinical Outcomes in Patients With Chronic Kidney Disease Undergoing Impella-Supported High-Risk Percutaneous Coronary Intervention: Insights From the cVAD PROTECT III Study. Circ Cardiovasc Interv. 2024 Jul;17(7):e013503. doi: 10.1161/CIRCINTERVENTIONS.123.013503. Epub 2024 May 6. PMID 38708609
- [Derived] Shah T, Abu-Much A, Batchelor WB, Grines CL, Baron SJ, Zhou Z, Li Y, Maini AS, Redfors B, Hussain Y, Wollmuth JR, Basir MB, O'Neill WW, Lansky AJ. Sex Differences in pLVAD-Assisted High-Risk Percutaneous Coronary Intervention: Insights From the PROTECT III Study. JACC Cardiovasc Interv. 2023 Jul 24;16(14):1721-1729. doi: 10.1016/j.jcin.2023.04.036. Epub 2023 Jul 5. PMID 37409991